CLINICAL TRIAL: NCT05809037
Title: Evaluation of Noninvasive Vagus Nerve Stimulation on Functional Status in Ischemic Stroke
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Istanbul Physical Medicine Rehabilitation Training and Research Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2022/382
Record Dates: First submitted 2023-03-30; First posted 2023-04-12 (Actual); Last update posted 2023-04-12 (Actual); Status verified 2023-04

CONDITIONS: Stroke, Ischemic; Hemiplegia; Hemiparesis;Poststroke/CVA
MeSH Terms: conditions — Ischemic Stroke; Hemiplegia

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Active Stimulation for right hemiparesis patients (Active Comparator): Active non-invasive transauricular vagus nerve stimulation over left ear in post-stroke right hemiparesis
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham Stimulation for right hemiparesis patients (Sham Comparator): Sham non-invasive transauricular vagus nerve stimulation over left ear in post-stroke right hemiparesis
  Interventions: Device: Sham stimulation
- Active Stimulation for left hemiparesis patients (Active Comparator): Active non-invasive transauricular vagus nerve stimulation over left ear in post-stroke left hemiparesis
  Interventions: Device: transcutaneous auricular vagus nerve stimulation
- Sham Stimulation for left hemiparesis patients (Sham Comparator): Sham non-invasive transauricular vagus nerve stimulation over left ear in post-stroke left hemiparesis
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: transcutaneous auricular vagus nerve stimulation — In addition to the conventional rehabilitation program, non-invasive vagus nerve stimulation will be applied to the participants through the left ear with the Vagustim™-Ear tens electrode. As a vagus stimulation protocol, 10 sessions, 30 minutes, noninvasive auricular stimulation will be applied, stimulation frequency is 10 Hz, pulse width is 300 µs, and biphasic.
  Arms: Active Stimulation for left hemiparesis patients; Active Stimulation for right hemiparesis patients
Device: Sham stimulation — In addition to the conventional rehabilitation program, sham vagus nerve stimulation (0 mA) will be applied to the participants in the control group. Non-invasive vagus nerve stimulation will be applied to the participants through the left ear with the Vagustim™-Ear tens electrode. As a vagus stimulation protocol, 10 sessions, 30 minutes, and noninvasive auricular stimulation will be applied.
  Arms: Sham Stimulation for left hemiparesis patients; Sham Stimulation for right hemiparesis patients

SUMMARY:
In this study, the effectiveness of vagus nerve stimulation in patients with right and left hemiparesis will be compared with each other and with the sham application.

DETAILED DESCRIPTION:
This prospective study will include 80 participants with a diagnosis of ischemic stroke who meet the inclusion criteria. In addition to the conventional rehabilitation program, non-invasive vagus nerve stimulation will be applied to the participants through the left ear with the Vagustim™-Ear tens electrode. As a vagus stimulation protocol, 10 sessions, 30 minutes, noninvasive auricular stimulation will be applied, stimulation frequency is 10 Hz, the pulse width is 300 µs, biphasic. In the study, sham vagus nerve stimulation (0 mA) will be applied to the participants in the control group. The study will be completed when the evaluation of the participants is made in the 1st and 3rd months after the last intervention. The upper extremity functions of the patients participating in the study were determined by Fugl-Meyer upper extremity test and box and block test, upper and lower extremity spasticities by modified Ashworth scale, and sleep quality by Pittsburgh sleep quality index. Quality of life will be evaluated with the stroke-specific quality of life scale, balance functions with the Berg balance test, dependency levels in daily activities with the Barthel index, and sympathetic dysfunctions with COMPASS-31. Participants' blood pressure and pulse values will be evaluated before and after each session.

ELIGIBILITY:
Inclusion Criteria:

* History of subacute-chronic ischemic stroke (3-12 months)

Exclusion Criteria:

* Bilateral or unilateral previous injury to the vagus nerve (eg injury during carotid endarterectomy).
* Severe depression (Beck Depression Scale > 29)
* Current use of any other stimulation device, such as a pacemaker or other neurostimulator; current use of any other investigational device or drug.
* Medical or mental instability (diagnosis of personality disorder, psychosis, or substance abuse) that would prevent the subject from following the protocol timeline.
* Pregnancy or planning to become pregnant or breastfeed during the study period.
* Botox injections or hemiplegia rehabilitation within 6 months before treatment.
* Having a history of hemorrhagic stroke
* Presence of ongoing dysphagia or aspiration difficulties.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-03-27 (Actual); Primary Completion 2023-12-27 (Estimated); Study Completion 2024-03-27 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment for Upper Extremity | Change from Baseline Fugl-Meyer Assessment for Upper Extremity at 4 weeks and 12 weeks
  It is considered as gold standard and is the only impairment level measure recommended for stroke trials. It consists of 30 items assessing motor function and 3 items assessing reflex function. The score most applicable to task performance is given from "0, inability," "1, beginning ability," to "2, normal" (total score range, 0-66).
Stroke-Specific Quality of Life Scale | Change from Baseline Stroke-Specific Quality of Life Scale at 4 weeks and 12 weeks
  The Stroke-Specific Quality of Life Scale assesses health-related quality of life specific to stroke survivors. 49 questions under 12 subscales. Scores range from 49-245. Higher scores indicate better functioning.

SECONDARY OUTCOMES:
Barthel Index | Change from Baseline Barthel Index at 4 weeks and 12 weeks
  Barthel Index is used to measure the disability experienced by the patient in performing activities of daily living. It comprises 10 items regarding activities of daily living and mobility and assesses feeding, transfer from wheelchair to bed and back, self-care, bathing, walking, climbing stairs, dressing, and bladder and bowel continence. Scoring is based on whether the patient requires help or not in performing any of the above mentioned activities. Proposed guidelines for interpreting Barthel scores are that scores of 0-20 indicate "total" dependency, 21-60 indicate "severe" dependency, 61-90 indicate "moderate" dependency, and 91-99 indicates "slight" dependency.
Modified Ashworth Scale | Change from Baseline Modified Ashworth Scale at 4 weeks and 12 weeks
  Modified Ashworth Scale (MAS) is used to assess spasticity. Scoring: 0: No increase in tone; 1: slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension; 1+: slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM ); 2: more marked increase in tone but more marked increased in muscle tone through most limb easily flexed; 3: considerable increase in tone, passive movement difficult and, 4: limb rigid in flexion or extension
Berg Balance Test | Change from Baseline Berg Balance Test at 4 weeks and 12 weeks
  Berg Balance Test is consisting of 14 items and measures the ability of individuals to maintain balance while performing functional tasks. Each task is scored from 0 (cannot perform independently) to 4 (stated best performance). 0-20 points are interpreted as high risk of falling, between 21-40 points as medium risk of falling, and between 41-56 points as low risk.
Composite Autonomic Symptom Score (COMPASS-31) | Change from Baseline Composite Autonomic Symptom Score at 4 weeks and 12 weeks
  The test has 6 domains looking at autonomic symptoms: orthostatic intolerance, vasomotor, secretomotor, gastrointestinal, bladder and pupillomotor. The six domain scores sum to a total COMPASS 31 score of 0 to 100, and a higher COMPASS 31 score indicates more severe autonomic symptoms.
Pittsburgh Sleep Quality Index | Change from Baseline Pittsburgh Sleep Quality Index at 4 weeks and 12 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-rated questionnaire which assesses sleep quality and disturbances over a 1-month time interval. Each item is weighted on a 0-3 interval scale. The global PSQI score is then calculated by totaling the seven component scores, providing an overall score ranging from 0 to 21, where lower scores denote a healthier sleep quality.

CONTACTS AND LOCATIONS:
Overall Officials: Selim Sezikli, MD, Principal Investigator — Istanbul Physical Medicine and Rehabilitation Training and Research Hospital
Locations (1):
- Istanbul Physical Medicine and Rehabilitation Training and research Hospital, Istanbul, Turkey (Türkiye)